CLINICAL TRIAL: NCT03828591
Title: The Impact of Psychological Support During the Hospitalization in Women With Endometriosis
Brief Title: Endometriosis and Psychological Support
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal Investigator, Renato Seracchioli, principal investigator, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ENDO.PS.
Record Dates: First submitted 2019-01-24; First posted 2019-02-04 (Actual); Last update posted 2019-05-15 (Actual); Status verified 2019-05

CONDITIONS: Endometriosis
Keywords: Endometriosis; Psychological support
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (intensive support) (Other): Patients that receive standard and intensive psychological support during hospitalization
  Interventions: Procedure: Intensive psychological support; Procedure: Standard psychological support
- Group B (standard support) (Other): Patients that receive only standard psychological support during hospitalization
  Interventions: Procedure: Standard psychological support

INTERVENTIONS:
Procedure: Intensive psychological support — Two meeting with a psychologist during the hospitalization (the first two days after surgery; the second one at the moment of the hospitalization discharge)
  Arms: Group A (intensive support)
Procedure: Standard psychological support — Two meetings with a psychologist: the first meeting is one month before surgery; the second meeting is one month after surgery

SUMMARY:
Endometriosis is a common disease, causing significant pain (dysmenorrhea, dysuria, dyspnea, dyspareunia, and chronic pelvic pain) and infertility, drastically reducing patients' quality of life.

Endometriosis surgery is often a stressful event for the patient. For that reason, psychological support can improve patients' general health state.

DETAILED DESCRIPTION:
Patients with clinical and trans-vaginal / abdominal ultrasound diagnosis of endometriosis, undergoing surgery for the removal of endometriotic lesions are included in the study.

Psychological support is offered to all women one month before and one month after surgery. A group of patients will receive intensive psychological support during hospitalization.

Patients are divided into 2 groups:

Group A: patients receiving intensive psychological support during hospitalization

Group B: patients not receiving intensive psychological support during hospitalization

After surgery, patients will be included in the post-operative follow-up, as usual in the investigator's clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing surgery for endometriosis
* Patients that have signed an informed consent

Exclusion Criteria:

* Patients with active or history of psychological/psychiatric diseases
* Patients that refuse psychological support

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-08 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
General health state | From one month before surgery until the hospitalization discharge; assessed up to 7 days after surgery
  Measurement of quality of life of patients underwent surgery for endometriosis, using the validated questionnaire Clinical Outcomes In Routine Evaluation, with a total score from 1 (the best outcome) to more than 85 (the worse outcome), where: 1 to 20 is Healthy; 21 to 33 is Low level; 34 to 50 is Mild level; 51 to 67 is Moderate level; 68 to 84 is Moderate to severe level; more than 85 is Severe level. The questionnaire is submitted one month before surgery and at the hospitalization discharge.

SECONDARY OUTCOMES:
Postoperative pain: Numeric Rating Scale | Postoperative: at the hospitalization discharge (assessed up to 7 days after surgery) and one month after surgery
  Evaluation of postoperative pain using Numeric Rating Scale, from 0 to 10 (where 0 is no pain and 10 is the worse pain ever).
Anxiety and Depression | From one month before surgery until the hospitalization discharge; assessed up to 7 days after surgery
  Measurement of anxiety and depression of patients underwent surgery for endometriosis, using the validated questionnaire Hospital Anxiety and Depression Scale, from 0 (the best outcome) to 21 (the worse outcome), where: 0 to 7 is Normal; 8 to 10 is Borderline case; 11 to 21 is Abnormal.
Stress | From one month before surgery until the hospitalization discharge; assessed up to 7 days after surgery
  Measurement of stress in patients underwent surgery for endometriosis, using the validated questionnaire Perceived Stress Scale, from 0 (the best outcome) to 40 (the worse outcome), where scores ranging from 0-13 would be considered low stress; scores ranging from 14-26 would be considered moderate stress; scores ranging from 27-40 would be considered high perceived stress.

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliero-Universitaria Sant'Orsola Malpighi, Bologna, BO, Italy